CLINICAL TRIAL: NCT03820011
Title: Feasibility Test of a Pediatric Web-Based Care Planning Guide
Brief Title: Participation and Environment Measure-Plus (PEM-Plus) Care Planning Intervention
Acronym: PEM-Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary A Khetani (Other)
Collaborators: McGill University (Other); McMaster University (Other)
Responsible Party: Sponsor-Investigator, Mary A Khetani, Associate Professor, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0600
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Developmental Disability; Early Intervention (Education)
Keywords: participation; environment; goal setting
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEM-Plus Group (Experimental): For Aim 1, 6 parents of young children were recruited to perform tasks related to navigating the PEM+ interface. Data on completion rate and time, as well as user satisfaction, were analyzed to guide PEM+ improvements. For Aim 2, we recruited 27 participants to enroll in a feasibility trial of PEM+. Caregivers who completed the YC-PEM e-PRO to evaluate their child's participation clicked on a weblink to begin PEM+, whereby they built on their YC-PEM responses for the purpose of creating a participation-focused care plan to share with their child's rehabilitation team. Caregivers were instructed to complete the PEM+ over a two-week (14 day) period because it mimics what would be provided in routine care.
  Interventions: Other: PEM+

INTERVENTIONS:
Other: PEM+ — PEM+ is a five-step recursive process (i.e., the caregiver can repeat the five-step process to create as many intervention plans for their child as needed, relative to the number of activities in which change is desired based on the YC-PEM e-PRO, and it offers tiered support to the user during completion (tier 1: frequently asked questions available in the application, tier 2: support provided by email, tier 3: support provided by phone).

SUMMARY:
The goal of the proposed research is to achieve a major advance in promoting effective and efficient delivery of pediatric rehabilitation services for young children with developmental disabilities and delays. The investigative team will examine the usability, feasibility, acceptability, and preliminary effects of PEM+, an innovative web-based (mobile friendly) guide for care planning by parents of young children with developmental disabilities and delays. PEM+ is designed in partnership with parents and providers to support more collaborative and efficient clinical care planning with individual families who typically access pediatric occupational therapy services. Specifically, PEM+ enables parents to build on their baseline assessment of their child using the Young Children's Participation and Environment Measure (YC-PEM) to design specific solutions to their young child's participation-related problems. PEM+ affords parents the opportunity to do this in their own space and on their own schedule, as well as electronically share their proposed written solutions with their child's provider(s) and/or other important individuals in their young child's life.

DETAILED DESCRIPTION:
Participation and Environment Measure Plus (PEM+) is a new electronic health application that facilitates family-centered and participation-focused intervention planning for young children receiving rehabilitation therapies. PEM+ design was informed by caregiver and provider input. It is a web-based intervention planning application that is designed for use by caregivers of young children receiving rehabilitation therapies. Caregivers who complete the Young Children's Participation and Environment Measure (YC-PEM), an electronic patient-reported outcome measure, evaluate their child's participation and then can click on a weblink to begin the PEM+ application, whereby they build on their YC-PEM responses for the purpose of creating a participation-focused care plan to share with their child's rehabilitation team. PEM+ is a five-step recursive process (i.e., the caregiver can repeat the five-step process to create as many care plans for their child as needed), and it offers tiered support to the user during completion (tier 1: frequently asked questions available in the application, tier 2: support provided by email, tier 3: support provided by phone). For the first aim of this study, caregivers completed one iteration of PEM+ to complete user tasks for the purpose of evaluating PEM+ usability. For the second aim of this study, caregivers were instructed to complete the PEM+ over a two-week (14 day) period. This time frame was selected by the research team as it mimics what would be provided in the routine care planning processes of early intervention and early childhood education.

ELIGIBILITY:
Aim 1 Inclusion Criteria:

* at least 18 years old
* reads, writes, and speaks English
* has access to broadband internet
* resides in the U.S
* has a child between 0 and 3 years old who is receiving services for developmental delay.

Aim 1 Exclusion Criteria:

* has a child over 3 years old
* does not have internet access
* has a child who is not receiving rehabilitation services for developmental delay
* does not reside in the U.S.

Aim 2 Inclusion Criteria:

* 18 years or older
* reads, writes, and speaks in English
* has a child aged 0-5 years old who was receiving rehabilitation services
* has broadband internet access
* denotes at least one area of desired change during participation assessment.

Aim 2 Exclusion Criteria:

* has a child over 5 years old
* does not have internet access
* has a child who is not receiving rehabilitation services for developmental delay
* does not reside in the U.S.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Khetani, ScD, Principal Investigator — Board of Trustees at University of Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PEM-Plus Group (Aim 1): For Aim 1, 6 parents of young children were recruited to perform tasks related to navigating the PEM+ interface during one iteration only. Data on completion rate and time, and user satisfaction, were analyzed to guide PEM+ improvements.
  PEM+ is a five-step recursive process, so the caregiver can repeat the five-step process to create as many intervention plans for their child as needed, and it offers tiered support.
- PEM-Plus Group (Aim 2): For Aim 2, we recruited 27 participants to enroll in a feasibility trial of PEM+. Caregivers who completed the YC-PEM e-PRO to evaluate their child's participation clicked on a weblink to begin PEM+, whereby they built on their YC-PEM responses for the purpose of creating a participation-focused care plan to share with their child's rehabilitation team. Caregivers were instructed to complete the PEM+ as many time as needed over a 14 day period because it mimics what would be provided in routine care.
  PEM+ is a five-step recursive process, so the caregiver can repeat the five-step process to create as many intervention plans for their child as needed, and it offers tiered support.
Period: Overall Study
Arm/Group | PEM-Plus Group (Aim 1) | PEM-Plus Group (Aim 2)
Started | 6 | 22
Completed | 6 | 18
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- PEM-Plus Group (Aim 2): For Aim 2, caregivers who completed the YC-PEM e-PRO clicked on a weblink to begin PEM+, whereby they built on their YC-PEM responses to create care plans to share with their child's rehabilitation team. Caregivers were instructed to complete the PEM+ over a 14-day period because it mimics routine care. PEM+ is a five-step recursive process (i.e., the caregiver repeats the process to create as many intervention plans for their child as needed), and it offers tiered support to the user during completion (tier 1: frequently asked questions available in the application, tier 2: support provided by email, tier 3: support provided by phone).
- PEM-Plus Group (Aim 1): For Aim 1, 6 parents of young children were recruited to perform tasks related to navigating the PEM+ interface. Data on completion rate and time and user satisfaction were analyzed to guide PEM+ improvements.
- Total: Total of all reporting groups
Arm/Group | PEM-Plus Group (Aim 2) | PEM-Plus Group (Aim 1) | Total
Number analyzed (Participants) | 22 | 6 | 28
Age, Categorical [Count of Participants; unit: Participants]
  Age of caregiver: <=18 years | 0 | 0 | 0
  Age of caregiver: Between 18 and 65 years | 22 | 6 | 28
  Age of caregiver: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 6 | 26
  Male | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 1 | 4
  Black or African American | 2 | 0 | 2
  White | 14 | 3 | 17
  Other or Not Disclosed | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Retention Rates
Description: As an indicator of PEM+ feasibility, we used web analytics to obtain estimates of the percentage of caregivers who enrolled completed the trial.
Time Frame: Following completion of two-week trial
Population: As stated in our published article, a total of 22 of the 27 participants recruited confirmed their eligibility, and 18 of the 22 participants who confirmed study eligibility continued with PEM+ use. This outcome is specific to Aim 2.
Measure: Count of Participants; unit: Participants
Arm/Group | PEM-Plus Group (Aim 2)
Number analyzed (Participants) | 22
Participants | 18

2. Primary Outcome: Median PEM+ Completion Time
Description: As an indicator of PEM+ feasibility, we used web analytics to estimate the median time for completing the first and subsequent iterations within a two-week trial period
Time Frame: Following completion of PEM+ iteration (Aim 1) and two weeks (Aim 2)
Measure: Median (Full Range); unit: minutes
Arm/Group | PEM-Plus Group (Aim 1) | PEM-Plus Group (Aim 2)
Number analyzed (Participants) | 6 | 18
minutes | 13.6 [3.3 to 20] | 12.99 [6.70 to 17.33]

3. Primary Outcome: Percentage of Caregivers Completing PEM+ Independently
Description: As an indicator of PEM+ feasibility, we used web analytics to estimate proportion of care plans created
Time Frame: Following completion of two-week trial
Measure: Count of Participants; unit: Participants
Arm/Group | PEM-Plus Group (Aim 2)
Number analyzed (Participants) | 18
Participants | 17

4. Primary Outcome: Median Number of PEM+ Care Plans Created
Description: As an indicator of PEM+ feasibility, we used web analytics estimate the number of care plans created over a two-week trial period.
Time Frame: Following completion of two-week trial
Population: This Outcome Measure was pre-specified to be only assessed under Aim 2 of the study. Aim 1 only required caregivers to complete a single iteration of PEM+, so all participants completed it one time. Aim 2 required caregivers to complete as many iterations of PEM+ as possible over 2 weeks, so participants could complete PEM+ one or more times.
Measure: Median (Full Range); unit: care plans
Arm/Group | PEM-Plus Group (Aim 2)
Number analyzed (Participants) | 18
care plans | 2.5 [1 to 17]

5. Primary Outcome: Usefulness, Satisfaction, and Ease of Use Questionnaire (USE)
Description: As an indicator of PEM+ acceptability, the USE is a questionnaire that evaluates usefulness, ease of use, ease of learning, and satisfaction. Items are on a 7-point scale, from from [1] strongly disagree, to [7] strongly agree. There were multiple items for each domain, which were summed together and divided by the total number of items to generate a summary score for that domain. Higher scores indicate a better outcome.
Time Frame: Following completion of two-week trial
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PEM-Plus Group (Aim 1): Aim 1 enrolled 6 caregivers to use PEM+ once and assess for its usability, results of which would inform optimizations prior to undertaking a Phase 1 trial.
Arm/Group | PEM-Plus Group (Aim 2) | PEM-Plus Group (Aim 1)
Number analyzed (Participants) | 18 | 6
score on a scale
  Usefulness | 4.41 (1.54) | NA (NA) — This domain of the USE outcome measure was not administered to decrease response burden, and it was deemed least relevance for Aim 1 targeting ease of use, learning, and satisfaction with an abbreviated intervention (i.e., one iteration).
  Ease of Use | 4.64 (1.25) | 4.4 (5.8)
  Ease of Learning | 4.97 (1.57) | 5.4 (6.0)
  Satisfaction | 3.80 (1.97) | 4.2 (5.7)

6. Primary Outcome: Caregiver Self-Efficacy to Promote Child's Participation in Activities
Description: As an indicator of preliminary effects, we developed two items for this project to estimate caregiver self-efficacy in caring for their child, according to "what I will do next [to support child's participation]" and "how I think [about my child's participation]". Each item was rated on a 7-point scale, from [1] strongly disagree, to [7] strongly agree. Higher scores indicate a better outcome.
Time Frame: Following completion of two-week trial
Population: This Outcome Measure was pre-specified to be only assessed under Aim 2 of the study, to identify clinical outcomes to include in a future efficacy trial of the PEM+ intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEM-Plus Group (Aim 2)
Number analyzed (Participants) | 18
score on a scale
  PEM+ influenced what I will do | 4.61 (1.85)
  PEM+ influenced what I think can be done | 4.72 (2.24)

ADVERSE EVENTS:
Time Frame: We collected data on adverse events for 10 months
Description: We did not report any adverse events in either Aim 1 or Aim 2 of this study.
Groups:
- PEM-Plus Group: For Aim 1, 6 parents of young children were recruited to perform tasks related to navigating the PEM+ interface during one iteration. Data on completion rate and time, and user satisfaction, were analyzed to guide PEM+ improvements. For Aim 2, we recruited 27 participants to enroll in a feasibility trial of PEM+. Caregivers who completed the YC-PEM e-PRO to evaluate their child's participation clicked on a weblink to begin PEM+, whereby they built on their YC-PEM responses to create a participation-focused care plan to share with their child's rehabilitation team. Caregivers were instructed to complete the PEM+ over a 14-day period because it mimics what would be provided in routine care. PEM+ is a five-step recursive process (i.e., the caregiver can repeat the five-step process to create as many intervention plans for their child as needed, and it offers tiered support to users).
Arm/Group | PEM-Plus Group
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
There were sampling limitations, as condition severity may impact PEM+ feasibility and the effect on caregiver confidence. There is a need to include a validated measure of caregiver confidence and/or self-efficacy in future PEM+ testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT03820011/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT03820011/SAP_001.pdf
  • Informed Consent Form (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03820011/ICF_002.pdf